CLINICAL TRIAL: NCT01318707
Title: Biomarkers Serum Collection Methodology Pilot Study
Status: Completed | Type: Observational
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Craig Kessler, IRB, Georgetown University
Other Study IDs: BiomarkersHemA
Record Dates: First submitted 2010-12-16; First posted 2011-03-18 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Hemophilia A
Keywords: Severe Hemophilia A; Hemophilia A Patients; Serum collection vs a method of added FVIII to blood samples
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare the standard collection of whole blood in tiger top tubes for serum collection versus a collection method of added FVIII to whole blood samples in the hemophilia population for routine biomarker assays to ensure reliable assay results.

DETAILED DESCRIPTION:
20 adults with severe Hemophilia A seen in one HTC site for routine blood drawing will be consented for discard blood sampling.

Half of the whole blood discard will be placed in a tiger top test tube, and half of the whole blood discard sample will be placed in a red top test tube containing exogenously added recombinant human FVIII concentrate [Advate, Baxter immuno] to assure an end concentration of once IU per CC of whole blood.

Both whole blood specimens will be allowed to coagulate at room temperature and then will be centrifuged to prepare serum. The separated serum from each type of collection test tubes will be aliquoted into eppendorf tubes (a minimum of two aliquots per sample) at a volume of 150 microliters. Aliquoted serum samples will be stored at -70 degrees centigrade and shipped on dry ice to Synarc Labs.

A panel of standard CTX bone resorption assays will be preformed in duplicate on the two differently processed serum specimens obtained from each subject.

Results will be analyzed for inter-subject variability using stored age-matched samples provided by Synarc and intra-subject variability will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Severe Hemophilia A

Exclusion Criteria:

* If they are not diagnosed with severe hemophilia A.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Severe Hemophilia A
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Kessler, MD, Principal Investigator — Georgetown University
Locations (1):
- Lombardi Cancer Center, Washington D.C., District of Columbia, United States